CLINICAL TRIAL: NCT01085331
Title: A Double-blind, Randomized, Comparative, Multicenter, Exploratory, and Placebo-controlled Phase II Trial of FOLFIRI Plus MSC1936369B or Placebo With a Safety run-in Part as Second-line Treatment of Metastatic K Ras Mutated Colorectal Cancer Subjects
Brief Title: MEK Inhibitor MSC1936369B Plus FOLFIRI in Second Line K-Ras Mutated Metastatic Colorectal Cancer (mCRC)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Conduct the randomized Phase 2 part not recommended due to the achieved MTD for pimasertib (45mg/day) in combination with FOLFIRI
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMR200066_004
Record Dates: First submitted 2010-03-04; First posted 2010-03-11 (Estimated); Results first posted 2016-10-19 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-08

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Mek Inhibitor; Metastatic Colorectal Cancer; K-Ras Mutation; Phase II; Second line K-Ras mutated metastatic colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — N-(2,3-dihydroxypropyl)-1-((2-fluoro-4-iodophenyl)amino)isonicotinamide; IFL protocol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1 or Safety Run-in Part: Pimasertib+FOLFIRI (Experimental)
  Interventions: Drug: Pimasertib; Drug: FOLFIRI
- Part 2 or Phase 2 Randomized part: Pimasertib+FOLFIRI (Experimental): Planned, not performed
  Interventions: Drug: Pimasertib; Drug: FOLFIRI
- Part 2 or Phase 2 Randomized part: Placebo+FOLFIRI (Experimental): Planned, not performed
  Interventions: Drug: Placebo; Drug: FOLFIRI

INTERVENTIONS:
Drug: Pimasertib — Subjects will be administered with pimasertib orally once daily on Days 1-5, 8-12, 15-19, and 22-26 of a 28 day cycle.
  Other Names: MSC1936369B
  Arms: Part 1 or Safety Run-in Part: Pimasertib+FOLFIRI; Part 2 or Phase 2 Randomized part: Pimasertib+FOLFIRI
Drug: Placebo — Subjects will be administered with placebo orally once daily on days 1-5, 8-12, 15-19, and 22-26 of a 28 day cycle.
  Arms: Part 2 or Phase 2 Randomized part: Placebo+FOLFIRI
Drug: FOLFIRI — Subjects will be administered with FOLFIRI (laevoleucovorin 200 milligram per square meter [mg/m^2] intravenous [i.v] infusion over 90 minutes or leucovorin [dl-leucovorin] 400 mg/m^2 i.v. infusion over 90 minutes; followed by irinotecan 180 mg/m^2 given as a 90-minute infusion in 500 milliliter [mL] dextrose 5%; followed by a bolus 5-fluorouracil [FU] 400 mg/m^2 and a 46-hour infusion 5-FU 2400 mg/m^2) at conventional doses on days 1 and 15 of the same 28 day cycle.

SUMMARY:
The research trial is testing the experimental treatment pimasertib (MSC1936369B) in combination with FOLFIRI, as second-line treatment in metastatic K Ras mutated colorectal cancer subjects. The study will be run in two parts:

Part 1, or Safety Run-in Part: Will determine the maximum tolerated dose and the recommended Phase 2 dose (RP2D) of pimasertib combined with FOLFIRI as second-line treatment in subjects with metastatic K Ras mutated colorectal cancer.

Part 2 or Phase 2 Randomised Part: Will assess the anti-tumor activity of pimasertib combined with FOLFIRI compared to FOLFIRI with placebo as second-line treatment in metastatic K Ras mutated colorectal cancer subjects.

Phase I which Is an open label dose escalation "3+3" cohort, non-randomized, safety Phase II which is a double blind randomized safety/efficacy

ELIGIBILITY:
Inclusion Criteria:

For Safety Run-in and Part 2 or Phase 2 Randomised Part

* Histologically confirmed K-Ras mutated colon/rectum cancer
* Subject's disease must have progressed during or after a first-line treatment for metastatic disease with oxaliplatin and fluoropyrimidines based chemotherapy with or without bevacizumab
* Evidence of metastatic measurable disease at trial entry as per Response Evaluation Criteria in Solid Tumors. Complete tumor assessment performed within 14 days prior to first trial drug administration
* Male/female subjects aged greater than or equal to (>=) 18 years
* Subject has read and understood the informed consent form
* Women of childbearing potential must have a negative blood pregnancy test at the screening visit. Subjects and their partners must be willing to avoid pregnancy during the trial

Exclusion Criteria:

For Safety Run-in and Part 2 or Phase 2 Randomised Part

* Bone marrow impairment
* Renal impairment
* Liver function and liver cell integrity abnormality
* History of central nervous system (CNS) metastases
* History of difficulty of swallowing, malabsorption or other chronic gastrointestinal disease
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) greater than (>)1
* Known human immunodeficiency virus (HIV) positivity, active hepatitis C, or active hepatitis B
* Has received extensive prior radiotherapy on more than 30 percent (%) of bone marrow reserves, or prior bone marrow/stem cell transplantation
* Has received chemotherapy, any investigational drug, or having participated in another clinical trial within the past 4 weeks prior to trial first drug administration
* Has a history of any other significant medical disease
* Past or current history (within the last 2 years prior to inclusion) of malignancies except for the indication under this study
* Has significant cardiac conduction abnormalities and/or pacemaker
* Is a pregnant or nursing female
* Has retinal degenerative disease, history of uveitis, or history of retinal vein occlusion
* Other significant disease that in the Investigator's opinion would exclude the subject from the trial
* Known hypersensitivity to the trial treatment(s) or diluents (when applicable), including placebo or other comparator drug(s)
* Legal incapacity or limited legal capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-03; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Serono S.A., Geneva
Locations (3):
- Research Site, Leuven, Belgium
- Research Site, Napoli, Italy
- Research Site, Barcelona, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First/last subject (informed consent): March 2010/September 2011. Last subject completed:May 2012.
Pre-assignment Details: Enrolled: 22 screened for eligibility; 6 were excluded (mainly non-fulfillment of inclusion or exclusion). 16 subjects were treated in a total of 4 centers (2 in Spain and 1 each in Belgium and Italy).
Groups:
- Part 1 or Safety Run-in Part: Pimasertib 45 mg +FOLFIRI: Pimasertib was administered orally at a dose of 45 milligrams per day (mg/day) once daily on Days 1-5, 8-12, 15-19, and 22-26 of a 28 day cycle along with FOLFIRI (laevoleucovorin 200 milligram per square meter [mg/m^2] intravenous [i.v] infusion over 90 minutes or leucovorin [dl-leucovorin] 400 mg/m^2 i.v. infusion over 90 minutes; followed by irinotecan 180 mg/m^2 given as a 90-minute infusion in 500 milliliter [mL] dextrose 5%; followed by a bolus 5-fluorouracil [FU] 400 mg/m^2 and a 46-hour infusion 5-FU 2400 mg/m^2.) at conventional doses on days 1 and 15 of the same 28 day cycle.
- Part 1 or Safety Run-in Part: Pimasertib 60 mg +FOLFIRI: Pimasertib was administered orally at a dose of 60 mg/day once daily on Days 1-5, 8-12, 15-19, and 22-26 of a 28 day cycle along with FOLFIRI (laevoleucovorin 200 milligram per square meter [mg/m^2] intravenous [i.v] infusion over 90 minutes or leucovorin [dl-leucovorin] 400 mg/m^2 i.v. infusion over 90 minutes; Irinotecan 180 mg/m^2 given as a 90-minute infusion in 500 milliliter [mL] dextrose 5%; followed by a bolus 5-fluorouracil [FU] 400 mg/m^2 and a 46-hour infusion 5-FU 2400 mg/m^2) at conventional doses on days 1 and 15 of the same 28 day cycle.
Period: Overall Study
Arm/Group | Part 1 or Safety Run-in Part: Pimasertib 45 mg +FOLFIRI | Part 1 or Safety Run-in Part: Pimasertib 60 mg +FOLFIRI
Started | 10 | 6
Completed | 10 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all subjects who received at least one (non-zero) administration of the trial medication (any of the 3 FOLFIRI drugs and pimasertib).
Groups:
- Part 1 or Safety Run-in Part: Pimasertib 45 mg +FOLFIRI: Pimasertib was administered orally at a dose of 45 mg/day once daily on Days 1-5, 8-12, 15-19, and 22-26 of a 28 day cycle along with FOLFIRI (laevoleucovorin 200 mg/m^2 i.v infusion over 90 minutes or leucovorin [dl-leucovorin] 400 mg/m^2 i.v. infusion over 90 minutes; followed by irinotecan 180 mg/m^2 given as a 90-minute infusion in 500 mL dextrose 5%; followed by a bolus 5-fluorouracil [FU] 400 mg/m^2 and a 46-hour infusion 5-FU 2400 mg/m^2) at conventional doses on days 1 and 15 of the same 28 day cycle.
- Part 1 or Safety Run-in Part: Pimasertib 60 mg +FOLFIRI: Pimasertib was administered orally at a dose of 60 mg/day once daily on Days 1-5, 8-12, 15-19, and 22-26 of a 28 day cycle along with FOLFIRI (laevoleucovorin 200 mg/m^2 i.v infusion over 90 minutes or leucovorin [dl-leucovorin] 400 mg/m^2 i.v. infusion over 90 minutes; followed by irinotecan 180 mg/m^2 given as a 90-minute infusion in 500 mL dextrose 5%; followed by a bolus 5-fluorouracil [FU] 400 mg/m^2 and a 46-hour infusion 5-FU 2400 mg/m^2) at conventional doses on days 1 and 15 of the same 28 day cycle.
- Total: Total of all reporting groups
Arm/Group | Part 1 or Safety Run-in Part: Pimasertib 45 mg +FOLFIRI | Part 1 or Safety Run-in Part: Pimasertib 60 mg +FOLFIRI | Total
Number analyzed (Participants) | 10 | 6 | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.3 (12.0) | 60.4 (17.2) | 61.6 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Part 1 or Safety Run-in Part: Maximum Tolerated Dose (MTD)
Description: MTD was defined as the dose level, at which the treatment-related dose limiting toxicity (DLT) occurred in >1 of 3 subjects or in >1 of 6 subjects. DLT was defined using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v3.0. Any Grade >=3 non-hematological toxicity except for Grade 4 asymptomatic increases in liver function tests (LFTs) reversible within 7 days in subjects with liver involvement, Grade 3 asymptomatic increases in LFTs reversible within 7 days in subjects without liver involvement, Grade 3 vomiting controlled with adequate and optimal therapy and prophylaxis, and Grade 3 diarrhea controlled with adequate and optimal anti-diarrhea therapy; any Grade 4 neutropenia lasing >5 days/ febrile neutropenia lasting >1 day; any Grade 4 thrombocytopenia/Grade 3 with bleeding; any treatment delay >2 weeks due to trial treatment-related adverse effects at any dose level and judged to be possibly or probably related to the trial treatment.
Time Frame: Baseline up to Day 28 (Part 1)
Population: as for baseline characteristics
Measure: Number; unit: mg
Groups:
- Pimasertib+FOLFIRI (Overall): Pimasertib was administered orally once daily 45 mg/day and 60 mg/day on Days 1-5, 8-12, 15-19, and 22-26 of a 28 day cycle along with FOLFIRI (laevoleucovorin 200 mg/m^2 i.v infusion over 90 minutes or leucovorin [dl-leucovorin] 400 mg/m^2 i.v. infusion over 90 minutes; followed by irinotecan 180 mg/m^2 given as a 90-minute infusion in 500 mL dextrose 5%; followed by a Bolus 5-fluorouracil [FU] 400 mg/m^2 and a 46-hour infusion 5-FU 2400 mg/m^2) at conventional doses on days 1 and 15 of the same 28 day cycle.
Arm/Group | Pimasertib+FOLFIRI (Overall)
Number analyzed (Participants) | 16
mg | 45

2. Primary Outcome: Part 2 or Phase 2 Randomised Part: Progression Free Survival (PFS)
Description: PFS was defined as time (in months) from the date of randomization to the first documentation of disease progression as reported and documented by the Investigator (i.e. radiological progression per RECIST v1.0) or death for any cause.
Time Frame: From randomization up to first documented disease progression maximum up to 2 years
Population: Part 2 or Phase 2 Randomized Part of the trial was not conducted. Hence, PFS was not evaluated for this study.
Groups:
- Part 2 or Phase 2 Randomized Part: Pimasertib+FOLFIRI: Pimasertib was to be administered orally once daily on Days 1-5, 8-12, 15-19, and 22-26 of a 28 day cycle along with FOLFIRI (laevoleucovorin 200 mg/m^2 i.v infusion over 90 minutes or leucovorin [dl-leucovorin] 400 mg/m^2 i.v. infusion over 90 minutes; followed by irinotecan 180 mg/m^2 as a 90-minute infusion in 500 mL dextrose 5%; followed by a bolus 5-fluorouracil [FU] 400 mg/m^2 and a 46-hour infusion 5-FU 2400 mg/m^2) at conventional doses on days 1 and 15 of the same 28 day cycle.
- Part 2 or Phase 2 Randomized Part: Placebo +FOLFIRI: Placebo was to be administered orally once daily on Days 1-5, 8-12, 15-19, and 22-26 of a 28 day cycle along with FOLFIRI (laevoleucovorin 200 mg/m^2 i.v infusion over 90 minutes or leucovorin [dl-leucovorin] 400 mg/m^2 i.v. infusion over 90 minutes; followed by irinotecan 180 mg/m^2 as a 90-minute infusion in 500 mL dextrose 5%; followed by a Bolus 5-fluorouracil [FU] 400 mg/m^2 and a 46-hour infusion 5-FU 2400 mg/m^2) at conventional doses on days 1 and 15 of the same 28 day cycle.
Arm/Group | Part 2 or Phase 2 Randomized Part: Pimasertib+FOLFIRI | Part 2 or Phase 2 Randomized Part: Placebo +FOLFIRI
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Part 1 or Safety Run-in Part: Number of Subjects With Treatment Emergent Adverse Events (TEAEs), Serious TEAEs, TEAEs Leading to Discontinuation and TEAEs Leading to Death
Description: An AE is defined as any new untoward medical occurrences/worsening of pre-existing medical condition without regard to possibility of causal relationship. An SAE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: From the first dose of study drug administration up to 28 days after the last dose of study drug administration
Population: as for baseline characteristics
Measure: Number; unit: Subjects
Arm/Group | Part 1 or Safety Run-in Part: Pimasertib 45 mg +FOLFIRI | Part 1 or Safety Run-in Part: Pimasertib 60 mg +FOLFIRI
Number analyzed (Participants) | 10 | 6
Subjects
  TEAE | 10 | 6
  Serious TEAE | 4 | 4
  TEAEs leading to discontinuation | 6 | 4
  TEAEs leading to death | 0 | 0

4. Secondary Outcome: Part 1 or Safety Run-in Part: Maximum Observed Plasma Concentration (Cmax) of Pimasertib, Irinotecan and SN-38
Time Frame: Day 1 and Day 8 for pimasertib; Day 1 and Day 15 for Irinotecan and SN-38
Population: The pharmacokinetic (PK) evaluation set included subjects who had an evaluable plasma concentration-time profile on any of the PK sampling days (Day 1 or 8 or 15). "n" signifies number of subjects evaluable in each category, respectively.
Measure: Median (Full Range); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part 1 or Safety Run-in Part: Pimasertib 45 mg +FOLFIRI | Part 1 or Safety Run-in Part: Pimasertib 60 mg +FOLFIRI
Number analyzed (Participants) | 10 | 6
nanogram per milliliter (ng/mL)
  Pimasertib: Day 1 (n=9, 6) | 145 [82.3 to 418] | 386 [163 to 516]
  Pimasertib: Day 8 (n=9, 6) | 196 [71.6 to 660] | 332 [214 to 638]
  Irinotecan: Day 1 (n=10, 6) | 2070 [1590 to 3060] | 1850 [1230 to 2110]
  Irinotecan: Day 15 (n=8, 6) | 2120 [1760 to 2840] | 1540 [1330 to 2420]
  SN-38: Day 1 (n=10, 6) | 20.4 [11.4 to 37.6] | 21.9 [15.8 to 46.3]
  SN-38: Day 15 (n=8, 6) | 15.1 [9.28 to 37.5] | 27 [9.31 to 51.2]

5. Secondary Outcome: Part 1 or Safety Run-in Part: Time to Reach Maximum Observed Concentration (Tmax) of Pimasertib, Irinotecan and SN-38
Time Frame: Day 1 and Day 8 for pimasertib; Day 1 and Day 15 for Irinotecan and SN-38
Population: as for outcome 4
Measure: Median (Full Range); unit: hour
Arm/Group | Part 1 or Safety Run-in Part: Pimasertib 45 mg +FOLFIRI | Part 1 or Safety Run-in Part: Pimasertib 60 mg +FOLFIRI
Number analyzed (Participants) | 10 | 6
hour
  Pimasertib: Day 1 (n=9, 6) | 2 [1.00 to 6.00] | 0.79 [0.50 to 4.00]
  Pimasertib: Day 8 (n=9, 6) | 1.5 [0.53 to 2.00] | 1.25 [0.50 to 2.50]
  Irinotecan: Day 1 (n=10, 6) | 1.5 [1.25 to 2.50] | 1.5 [1.50 to 2.50]
  Irinotecan: Day 15 (n=8, 6) | 1.54 [1.50 to 2.50] | 1.56 [1.50 to 4.00]
  SN-38: Day 1 (n=10, 6) | 1.5 [1.50 to 2.25] | 1.5 [1.50 to 4.00]
  SN-38: Day 15 (n=8, 6) | 1.6 [1.50 to 2.50] | 2.5 [1.50 to 4.33]

6. Secondary Outcome: Part 1 or Safety Run-in Part: Area Under the Concentration-time Curve From Time Zero to the Time of Last Observation (AUC0-t) of Pimasertib, Irinotecan and SN-38
Description: Area under the plasma concentration-time curve from time zero to the last sampling time (AUC0-t) at which the concentration is at or above the lower limit of quantification.
Time Frame: Day 1 and Day 8 for pimasertib; Day 1 and Day 15 for Irinotecan and SN-38
Population: as for outcome 4
Measure: Median (Full Range); unit: (nanogram/milliliter)*hour([ng/mL]*hour)
Arm/Group | Part 1 or Safety Run-in Part: Pimasertib 45 mg +FOLFIRI | Part 1 or Safety Run-in Part: Pimasertib 60 mg +FOLFIRI
Number analyzed (Participants) | 10 | 6
(nanogram/milliliter)*hour([ng/mL]*hour)
  Pimasertib: Day 1 (n=9, 5) | 1120 [194 to 1860] | 1390 [666 to 2190]
  Pimasertib: Day 8 (n=8, 5) | 1270 [190 to 2030] | 1260 [858 to 2060]
  Irinotecan: Day 1 (n=10, 6) | 10500 [7130 to 18500] | 10200 [6220 to 11300]
  Irinotecan: Day 15 (n=8, 6) | 12700 [7040 to 17900] | 11400 [7050 to 13400]
  SN-38: Day 1 (n=10, 6) | 10500 [7130 to 18500] | 10200 [6220 to 11300]
  SN-38: Day 15 (n=8, 6) | 12700 [7040 to 17900] | 11400 [7050 to 13400]

7. Secondary Outcome: Part 1 or Safety Run-in Part: Area Under the Concentration-time Curve From Time Zero to Infinity (AUC0-inf) of Pimasertib, Irinotecan and SN-38
Description: The AUC(0-inf) of pimasertib and irinotecan was estimated by determining the total area under the concentration time curve extrapolated to infinity.
Time Frame: Day 1 and Day 8 for pimasertib; Day 1 and Day 15 for Irinotecan and SN-38
Population: The PK analysis population set included all subjects who had an evaluable plasma concentration-time profile on any of the PK sampling days (Day 1 or 8 or 15). Here, N (total number of subjects analyzed) signifies number of evaluable subjects for this outcome measure. "n" signifies number of subjects evaluable per each category, respectively.
Measure: Median (Full Range); unit: ng/mL*hour
Arm/Group | Part 1 or Safety Run-in Part: Pimasertib 45 mg +FOLFIRI | Part 1 or Safety Run-in Part: Pimasertib 60 mg +FOLFIRI
Number analyzed (Participants) | 9 | 6
ng/mL*hour
  Pimasertib: Day 1 (n=7, 5) | 1160 [226 to 1950] | 1430 [673 to 2310]
  Pimasertib: Day 8 (n=8, 5) | 1340 [244 to 2140] | 1340 [869 to 2170]
  Irinotecan: Day 1 (n=9, 6) | 10600 [7650 to 20600] | 11200 [6560 to 12500]
  Irinotecan: Day 15 (n=8, 6) | 13600 [7330 to 20400] | 12300 [7520 to 14500]
  SN-38: Day 1 (n=9, 6) | 10600 [7650 to 20600] | 11200 [6560 to 12500]
  SN-38: Day 15 (n=8, 6) | 13600 [7330 to 20400] | 12300 [7520 to 14500]

8. Secondary Outcome: Part 1 or Safety Run-in Part: Apparent Terminal Half Life (t1/2) of Pimasertib, Irinotecan and SN-38
Description: The t1/2 was defined as the time required for the plasma concentration of pimasertib and irinotecan to decrease 50% in the final stage of elimination.
Time Frame: Day 1 and Day 8 for pimasertib; Day 1 and Day 15 for Irinotecan and SN-38
Population: as for outcome 7
Measure: Median (Full Range); unit: hour
Arm/Group | Part 1 or Safety Run-in Part: Pimasertib 45 mg +FOLFIRI | Part 1 or Safety Run-in Part: Pimasertib 60 mg +FOLFIRI
Number analyzed (Participants) | 9 | 6
hour
  Pimasertib: Day 1 (n=7, 5) | 5.31 [2.37 to 5.97] | 5.56 [3.53 to 6.56]
  Pimasertib: Day 8 (n=8, 5) | 5.12 [3.88 to 7.27] | 5.08 [4.27 to 6.25]
  Irinotecan: Day 1 (n=9, 6) | 6.43 [5.32 to 7.63] | 6.83 [5.46 to 7.85]
  Irinotecan: Day 15 (n=8, 6) | 6.21 [5.54 to 8.77] | 6.45 [5.59 to 7.21]
  SN-38: Day 1 (n=9, 6) | 6.43 [5.32 to 7.63] | 6.83 [5.46 to 7.85]
  SN-38: Day 15 (n=8, 6) | 6.21 [5.54 to 8.77] | 6.45 [5.59 to 7.21]

9. Secondary Outcome: Part 1 or Safety Run-in Part: Apparent Oral Clearance (CL/f) of Pimasertib, (CL) Irinotecan and SN-38
Description: Clearance of a drug was a measure of the rate at which drug was metabolized or eliminated by normal biological processes. Apparent clearance after oral dose (CL/f) is influenced by the fraction absorbed.
Time Frame: Day 1 and Day 8 for pimasertib; Day 1 and Day 15 for Irinotecan and SN-38
Population: as for outcome 7
Measure: Median (Full Range); unit: Liter per hour
Arm/Group | Part 1 or Safety Run-in Part: Pimasertib 45 mg +FOLFIRI | Part 1 or Safety Run-in Part: Pimasertib 60 mg +FOLFIRI
Number analyzed (Participants) | 9 | 6
Liter per hour
  Pimasertib: Day 1 (n=7, 5) | 38.7 [23.1 to 199] | 42.1 [25.9 to 89.1]
  Pimasertib: Day 8 (n=8, 5) | 34.2 [21.0 to 184] | 44.6 [27.6 to 69.1]
  Irinotecan: Day 1 (n=9, 6) | 29.4 [16.4 to 47.0] | 29.7 [25.9 to 42.7]
  Irinotecan: Day 15 (n=8, 6) | 23.5 [15.6 to 46.8] | 26.2 [20.9 to 37.3]
  SN-38: Day 1 (n=9, 6) | 29.4 [16.4 to 47.0] | 29.7 [25.9 to 42.7]
  SN-38: Day 15 (n=8, 6) | 23.5 [15.6 to 46.8] | 26.2 [20.9 to 37.3]

10. Secondary Outcome: Part 1 or Safety Run-in Part: Apparent Oral Volume of Distribution (Vz f) Pimasertib, (Vz) of Irinotecan and SN-38
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired serum concentration. Apparent volume of distribution after oral dose (Vz/f) was influenced by the fraction absorbed.
Time Frame: Day 1 and Day 8 for pimasertib; Day 1 and Day 15 for Irinotecan and SN-38
Population: as for outcome 7
Measure: Median (Full Range); unit: Liter
Arm/Group | Part 1 or Safety Run-in Part: Pimasertib 45 mg +FOLFIRI | Part 1 or Safety Run-in Part: Pimasertib 60 mg +FOLFIRI
Number analyzed (Participants) | 9 | 6
Liter
  Pimasertib: Day 1 (n=7, 5) | 276 [197 to 680] | 348 [210 to 570]
  Pimasertib: Day 8 (n=8, 5) | 265 [189 to 1030] | 395 [246 to 425]
  Irinotecan: Day 1 (n=9, 6) | 297 [147 to 455] | 313 [241 to 395]
  Irinotecan: Day 15 (n=8, 6) | 212 [143 to 382] | 253 [182 to 336]
  SN-38: Day 1 (n=9, 6) | 297 [147 to 455] | 313 [241 to 395]
  SN-38: Day 15 (n=8, 6) | 212 [143 to 382] | 253 [182 to 336]

11. Secondary Outcome: Part 1 or Safety Run-in Part: Ratio of Cmax for Pimasertib (Day 1/Day 8), Irinotecan and SN-38 (Day 1/Day 15)
Time Frame: Day 1 and Day 8 for pimasertib; Day 1 and Day 15 for Irinotecan and SN-38
Population: as for outcome 7
Measure: Median (Full Range); unit: Ratio of Cmax
Arm/Group | Part 1 or Safety Run-in Part: Pimasertib 45 mg +FOLFIRI | Part 1 or Safety Run-in Part: Pimasertib 60 mg +FOLFIRI
Number analyzed (Participants) | 8 | 6
Ratio of Cmax
  Pimasertib (n=8, 5) | 0.837 [0.345 to 1.18] | 0.751 [0.359 to 2.22]
  Irinotecan (n=8, 6) | 0.973 [0.623 to 1.13] | 1.09 [0.774 to 1.40]
  SN-38 (n=8, 6) | 0.973 [0.623 to 1.13] | 1.09 [0.774 to 1.40]

12. Secondary Outcome: Part 1 or Safety Run-in Part: Ratio of AUC0-inf of Pimasertib (Day 1/Day 8), Irinotecan and SN-38 (Day 1/Day 15)
Description: The AUC(0-inf) was estimated by determining the total area under the concentration time curve extrapolated to infinity.
Time Frame: Day 1 and Day 8 for pimasertib; Day 1 and Day 15 for Irinotecan
Population: as for outcome 7
Measure: Median (Full Range); unit: Ratio
Arm/Group | Part 1 or Safety Run-in Part: Pimasertib 45 mg +FOLFIRI | Part 1 or Safety Run-in Part: Pimasertib 60 mg +FOLFIRI
Number analyzed (Participants) | 8 | 6
Ratio
  Pimasertib (n=7, 4) | 0.917 [0.738 to 1.22] | 0.825 [0.759 to 1.21]
  Irinotecan (n=8, 6) | 0.911 [0.577 to 1.08] | 0.844 [0.697 to 1.17]
  SN-38 (n=8, 6) | 0.911 [0.577 to 1.08] | 0.844 [0.697 to 1.17]

13. Secondary Outcome: Part 1 or Safety Run-in Part: Number of Subjects With Best Overall Response (BOR)
Description: BOR was defined based on Response Evaluation Criteria in Solid Tumors Version 1.0 (RECIST V1.0) as following: Complete response (CR) was defined as the disappearance of all target and non-target lesions and no appearance of new lesions. Partial response (PR) was defined as at least a 30 percent (%) decrease in the sum of the longest diameters (SLD) of the targeted lesions. CR and PR had to be documented on 2 occasions separated by at least 4 weeks (28 days). Stable disease (SD) was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify as progressive disease (PD) being demonstrated during the first 4 weeks. PD was defined as at least a 20% increase in the SLD of target lesions compared to the smallest SLD since the study treatment started.
Time Frame: Up to 2 years
Population: The efficacy analysis set included all subjects who received at least 1 trial drug dose (any of the three FOLFIRI drugs and pimasertib) and had a baseline tumor assessment and at least 1 post-baseline efficacy assessment.
Measure: Number; unit: Subjects
Arm/Group | Part 1 or Safety Run-in Part: Pimasertib 45 mg +FOLFIRI | Part 1 or Safety Run-in Part: Pimasertib 60 mg +FOLFIRI
Number analyzed (Participants) | 9 | 6
Subjects
  CR | 0 | 0
  PR | 1 | 1
  SD | 6 | 3
  PD | 1 | 2
  Not evaluable | 1 | 0

14. Secondary Outcome: Part 1 or Safety Run-in Part: Circulating Biomarkers in Serum
Time Frame: Predose, Day 1, 2 and 16 of cycle 1 followed by Day 1 pre-dose of every second cycle up to 2 years
Population: Number of subjects enrolled in the safety run-in part of the trial was less and it would not provide sufficient statistical power to perform any analysis. Hence, the biomarker samples were not analyzed as part of the trial.
Arm/Group | Part 1 or Safety Run-in Part: Pimasertib 45 mg +FOLFIRI | Part 1 or Safety Run-in Part: Pimasertib 60 mg +FOLFIRI
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Part 2 or Phase 2 Randomized Part: Circulating Biomarkers
Time Frame: Predose, Day 1, 2 and 16 of cycle 1 followed by Day 1 pre-dose of every second cycle up to 2 years
Population: Part 2 or Phase 2 Randomized Part of the trial was not conducted. Hence, circulating biomarkers were not evaluated.
Groups:
- Part 2 or Phase 2 Randomized Part: Placebo+FOLFIRI: Placebo was to be administered orally once daily on Days 1-5, 8-12, 15-19, and 22-26 of a 28 day cycle along with FOLFIRI (laevoleucovorin 200 mg/m^2 i.v infusion over 90 minutes or leucovorin [dl-leucovorin] 400 mg/m^2 i.v. infusion over 90 minutes; followed by irinotecan 180 mg/m^2 as a 90-minute infusion in 500 mL dextrose 5%; followed by a bolus 5-fluorouracil [FU] 400 mg/m^2 and a 46-hour infusion 5-FU 2400 mg/m^2) at conventional doses on days 1 and 15 of the same 28 day cycle.
Arm/Group | Part 2 or Phase 2 Randomized Part: Pimasertib+FOLFIRI | Part 2 or Phase 2 Randomized Part: Placebo+FOLFIRI
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Part 2 or Phase 2 Randomized Part: Best Overall Response
Description: as for outcome 13
Time Frame: Up to 2 years
Population: Part 2 or Phase 2 Randomized Part of the trial was not conducted. Hence, Best overall response was not evaluated.
Arm/Group | Part 2 or Phase 2 Randomized Part: Pimasertib+FOLFIRI | Part 2 or Phase 2 Randomized Part: Placebo+FOLFIRI
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Part 2 or Phase 2 Randomized Part: Number of Subjects With TEAEs, Serious TEAEs, TEAEs Leading to Discontinuation and TEAEs Leading to Death
Description: An AE is defined as any new untoward medical occurrences/worsening of pre-existing medical condition without regard to possibility of causal relationship. An SAE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect. TEAES between first dose of study drug administration and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: From the first dose of study drug administration up to 28 days after the last dose of study drug administration
Population: Part 2 or Phase 2 Randomized Part of the trial was not conducted. Hence, safety outcome measure could not be performed.
Arm/Group | Part 2 or Phase 2 Randomized Part: Pimasertib+FOLFIRI | Part 2 or Phase 2 Randomized Part: Placebo+FOLFIRI
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study drug administration up to 28 days after the last dose of study drug administration.
Arm/Group | Part 1 or Safety Run-in Part: Pimasertib 45 mg +FOLFIRI | Part 1 or Safety Run-in Part: Pimasertib 60 mg +FOLFIRI
Serious Adverse Events (participants affected / at risk) | 4/10 | 4/6
Other Adverse Events (participants affected / at risk) | 10/10 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 or Safety Run-in Part: Pimasertib 45 mg +FOLFIRI (N=10) | Part 1 or Safety Run-in Part: Pimasertib 60 mg +FOLFIRI (N=6)
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Mucosal inflammation (General disorders) | 0 | 2
Asthenia (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 0
Perirectal abscess (Infections and infestations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 or Safety Run-in Part: Pimasertib 45 mg +FOLFIRI (N=10) | Part 1 or Safety Run-in Part: Pimasertib 60 mg +FOLFIRI (N=6)
Asthenia (General disorders) | 6 | 4
Diarrhoea (Gastrointestinal disorders) | 8 | 5
Nausea (Gastrointestinal disorders) | 5 | 3
Vomiting (Gastrointestinal disorders) | 4 | 4
Stomatitis (Gastrointestinal disorders) | 2 | 5
Abdominal pain (Gastrointestinal disorders) | 3 | 3
Constipation (Gastrointestinal disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0
Mucosal inflammation (General disorders) | 3 | 2
Pyrexia (General disorders) | 3 | 2
fatigue (General disorders) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 4 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 4
Anaemia (Blood and lymphatic system disorders) | 3 | 0
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 1
Dizziness (Nervous system disorders) | 1 | 1
Dysgeusia (Nervous system disorders) | 1 | 1
Neurotoxicity (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Visual field defect (Nervous system disorders) | 1 | 0
Detachment of retinal pigment epithelium (Eye disorders) | 3 | 0
Macular degeneration (Eye disorders) | 2 | 1
Maculopathy (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Rash pustular (Infections and infestations) | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Electrocardiogram T wave inversion (Investigations) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Faecaluria (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal pain (Renal and urinary disorders) | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Procedural site reaction (Injury, poisoning and procedural complications) | 1 | 0
Depressed mood (Psychiatric disorders) | 1 | 0
Embolism (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
During the trial, the decision was made not to perform the Phase 2 part of the study due to the achieved MTD for pimasertib (45mg/day) in combination with FOLFIRI, so that no further dose escalation was possible as per the protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other